CLINICAL TRIAL: NCT04901611
Title: A Randomised Controlled Trial to Investigate the Effects of Parental Touch on Relieving Acute Procedural Pain in Neonates
Brief Title: Parental Touch Trial (Petal)
Acronym: Petal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paediatric Neuroimaging Research Group (Other)
Collaborators: Wellcome Trust (Other); University of Oxford (Other); Bliss Charity (Other)
Responsible Party: Principal Investigator, Rebeccah Slater, Professor of Paediatric Neuroscience, Paediatric Neuroimaging Research Group
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Petal
Record Dates: First submitted 2021-05-13; First posted 2021-05-25 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Infant Development; Pain, Procedural; Parents
Keywords: Parental touch; Brain activity; Stroking; Anxiety; Clinical pain score; Heart rate; Respiratory rate
MeSH Terms: conditions — Pain, Procedural; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parental touch (pre-procedural) (Experimental): Parents will stroke their baby on the posterior lower limb of the leg where the heel lance will be administered, at a speed of 3cm/s for 10 seconds using the whole hand and in one direction down the limb towards the foot. This will happen just before the control procedure and clinical heel lance.
  Interventions: Behavioral: Parental touch
- Parental touch (post-procedural) (Placebo Comparator): Parents will stroke their baby on the posterior lower limb of the leg where the heel lance was administered, at a speed of 3cm/s for 10 seconds using the whole hand and in one direction down the limb towards the foot. This will happen just after the control procedure and clinical heel lance.
  Interventions: Behavioral: Parental touch

INTERVENTIONS:
Behavioral: Parental touch — Parental touch in the form of stroking at 3cm/s for 10 seconds on the posterior lower limb where the heel lance will be/has been administered

SUMMARY:
This is a two centre two-arm randomised controlled interventional trial. We aim to determine whether parental touch prior to a painful clinical procedure provides effective analgesia in neonates.

DETAILED DESCRIPTION:
This is a multicentre randomised-controlled interventional trial, with two research sites (John Radcliffe Hospital, Oxford, and Royal Devon and Royal Devon and Exeter Hospital, Devon). In this study we aim to determine whether parental touch prior to a painful clinical procedure provides effective analgesia.

The primary objective is to determine whether parental touch reduces noxious-evoked brain activity following a heel lance. In addition, our secondary and exploratory objectives include investigating the effect of touch on behavioural and electrophysiological measures evoked by a heel lance. Neonates will be randomised to receive parental touch either prior to or post a clinically required heel lance. We will also investigate how parental touch impacts post-procedural clinical stability and explore whether this intervention affects parental anxiety.

Neonates will be recruited during a 9-month period. Participants will be studied on a single test occasion while they are in hospital, when they require a clinical heel lance. No extra blood tests or noxious procedures will be performed for the purpose of the study. Participants will be included in the study for approximately an hour period. This will be approximately 30 min before and after the time when the heel lance is performed. Individual babies will only be included in the trial once. If a neonate requires additional heel lances to acquire sufficient blood for clinical assessment at the time of the test occasion, we will also record the responses to this.

ELIGIBILITY:
Inclusion Criteria:

* Participants born at the John Radcliffe Hospital, Oxford or the Royal Devon and Exeter Hospital, Devon
* Neonates born at or after 35+0 weeks gestation
* Neonates with a postnatal age of 7 days or less
* Neonates who clinically require a heel lance
* Neonates for whom parents/guardians have given written informed consent for inclusion in the trial

Exclusion Criteria:

* Intraventricular haemorrhage (IVH) > grade II
* Received any analgesics or sedatives in the last 24 hours
* Congenital malformation or genetic condition known to affect neurological development
* Born to mothers who have a history of substance abuse.

Ages: 0 Days to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Magnitude of noxious-evoked brain activity | Immediately after heel lance (within 1000ms)
  An electroencephalography (EEG) template based on the Principal Component that reflects the noxious-evoked brain activity in neonates has been defined and validated in independent data sets (Hartley 2017). This template will be projected onto the EEG data recorded in the 1000ms period following each heel lance and heel lance control stimulus and the relative weight of the component calculated for each neonate. A greater weight indicates a stronger noxious-evoked response.

SECONDARY OUTCOMES:
Premature Infant Pain Profile - Revised score (PIPP-R score) | During the 30s period after the heel lance
  PIPP-R is a composite measure encompassing behavioural, physiological and contextual indicators involved in the pain response. These include gestational age, behavioural state, heart rate, oxygen saturation, and duration of brow bulge, eye squeeze, and nasolabial furrow. Each indicator in the PIPP-R is rated on a 4-point scale (0, 1, 2, and 3); these are summed together to produce a maximum possible score of 21, and minimum possible score of 0. In the revised PIPP-R, the scores for the contextual indicators (gestational age and behavioural state) are only included if a non-zero score is recorded for either the physiological or behavioural variables (Stevens et al., 2014). A higher score suggests a greater pain response.
Percentage of neonates who develop tachycardia | During the 30s period after the heel lance
  Percentage of neonates who develop post-procedural tachycardia (in the 30 seconds post-heel lance). Tachycardia will be defined as a heart rate >160 beats per minute as per Advanced Paediatric Life Support guidelines, reflecting heart rate values >90th centile for newborns in the first week of life (Fleming et al., 2011; Schwartz et al., 2002).
Parental anxiety | At the end of the test occasion, within 30 minutes of the heel lance
  Anxiety score from the 20-point Stait Trait Anxiety Inventory (STAI), the gold standard for state anxiety. It is well validated and publicly available. The STAI has a trait (STAI-T) and a state version (STAI-S). The STAI-T scale consists of 20 statements that ask people to describe how they generally feel. The STAI-S scale also consists of 20 statements, but the instructions require subjects to indicate how they feel at a particular moment in time. The STAI-S scale can be used to determine the actual levels of anxiety intensity induced by stressful procedures. Each question is rated on a 4-point scale (not at all, somewhat, moderately so, very much so). The range of possible scores for form Y of the STAI varies from a minimum score of 20 to a maximum score of 80 on both the STAI-T and STAI-S subscales. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).

OTHER OUTCOMES:
Exploratory outcome: changes in brain activity during parental touch intervention | During parental touch intervention
  Changes in brain activity recorded using EEG, which are elicited during the parental touch intervention. This is an exploratory outcome, therefore data will be investigated with a pragmatic approach.
Exploratory outcome: time taken for heart rate to return to baseline post-heel lance | 30 min time period after the clinical heel lance
  Impact of parental touch prior to the clinical procedure on reducing the duration of time for heart rate to return to baseline after a clinically-essential heel lance, compared with post-procedural touch.
Exploratory outcome: post-procedural variability in respiratory rate, incidence of apnoea, and change in respiratory stability | 30 min time period after the clinical heel lance
  Changes in respiratory rate and respiratory stability recorded using electrocardiogram (ECG). The data will also identify incidence of apnoea; an episode of apnoea will be defined as the cessation in breathing for at least 20s. This is an exploratory outcome, therefore data will be investigated with a pragmatic approach. Variability in respiratory rate, incidence of apnoea and change in respiratory stability are considered as one exploratory outcome as they are recorded using the same measurement techniques and interrelated.
Exploratory outcome: parental views | At the end of the test occasion, within 30 minutes of the heel lance
  Scores for each emotion, experienced by the parent during the heel lance, using a 4-point distress score (worried/upset/anxious/sad), and responses to a questionnaire about participating in this study and general infant research.

CONTACTS AND LOCATIONS:
Overall Officials: Eleri Adams, Principal Investigator — Oxford University Hospitals NHS Trust; Ravi Poorun, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the PI (rebeccah.slater@paediatrics.ox.ac.uk) listed on clinicaltrials.gov. The Study Protocol, Informed Consent Form and Statistical Analysis Plan will be available to download as a supplement to the final publication of the results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available after the publication of final results.
Access Criteria: PI will have discretion to share data with potential collaborators.

REFERENCES:
- [Derived] Baxter L, Hauck AGV, Bhatt A, Cobo MM, Hartley C, Marchant S, Poorun R, van der Vaart M, Slater R. Statistical analysis plan for the Petal trial: the effects of parental touch on relieving acute procedural pain in neonates. Wellcome Open Res. 2024 Dec 18;8:402. doi: 10.12688/wellcomeopenres.19819.3. eCollection 2023. PMID 40110538
- [Derived] Hauck AGV, van der Vaart M, Adams E, Baxter L, Bhatt A, Crankshaw D, Dhami A, Evans Fry R, Freire MBO, Hartley C, Mansfield RC, Marchant S, Monk V, Moultrie F, Peck M, Robinson S, Yong J, Poorun R, Cobo MM, Slater R. Effect of parental touch on relieving acute procedural pain in neonates and parental anxiety (Petal): a multicentre, randomised controlled trial in the UK. Lancet Child Adolesc Health. 2024 Apr;8(4):259-269. doi: 10.1016/S2352-4642(23)00340-1. Epub 2024 Feb 16. PMID 38373429
- [Derived] van der Vaart M, Hauck AGV, Mansfield R, Adams E, Bhatt A, Cobo MM, Crankshaw D, Dhami A, Hartley C, Monk V, Evans Fry R, Moultrie F, Robinson S, Yong J, Poorun R, Baxter L, Slater R. Parental experience of neonatal pain research while participating in the Parental touch trial (Petal). Pain. 2024 Aug 1;165(8):1727-1734. doi: 10.1097/j.pain.0000000000003177. Epub 2024 Jan 25. PMID 38284396
- [Derived] Cobo MM, Moultrie F, Hauck AGV, Crankshaw D, Monk V, Hartley C, Evans Fry R, Robinson S, van der Vaart M, Baxter L, Adams E, Poorun R, Bhatt A, Slater R. Multicentre, randomised controlled trial to investigate the effects of parental touch on relieving acute procedural pain in neonates (Petal). BMJ Open. 2022 Jul 19;12(7):e061841. doi: 10.1136/bmjopen-2022-061841. PMID 36250332